CLINICAL TRIAL: NCT06554171
Title: Investigation of the Effect of Hippotherapy Simulators on Trunk Control and Upper Extremity Functions in Children With Cerebral Palsy
Brief Title: Hippotherapy Simulators on Trunk Control and Upper Extremity Functions in Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/10-03
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Hippotherapy smilator; Upper extremity
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hippotherapy group (Experimental): In addition to conventional physiotherapy, training will be given in the Hippotherapy Simulator for 15 minutes a day, 5 days a week for 4 weeks. The hippotherapy simulator serves a wide range of purposes from recreational use that mimics the movements of a real horse or can make similar movements, to fitness, exercise, sports, education and therapy and is suitable for use by individuals with cerebral palsy.
  Interventions: Other: Hippotherapy group
- Control group (Experimental): In addition to conventional physiotherapy, the control group will be allowed to sit in the Hippotherapy Simulature for 15 minutes a day, 5 days a week for 4 weeks. However, the simulator will be kept in closed position to prevent oscillations.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Hippotherapy group — In addition to conventional physiotherapy, training will be given in the Hippotherapy Simulator for 15 minutes a day, 5 days a week for 4 weeks. The hippotherapy simulator serves a wide range of purposes from recreational use that mimics the movements of a real horse or can make similar movements, to fitness, exercise, sports, education and therapy and is suitable for use by individuals with cerebral palsy.
  Arms: Hippotherapy group
Other: Control group — In addition to conventional physiotherapy, the control group will be allowed to sit in the Hippotherapy Simulature for 15 minutes a day, 5 days a week for 4 weeks. However, the simulator will be kept in closed position to prevent oscillations.
  Arms: Control group

SUMMARY:
The hippotherapy simulator imitates the three-dimensional mechanical movement and walking of the horse and transfers the mechanical effect to the rider during hippotherapy. The aim of this study was to investigate the effect of exercise program with hippotherapy simulator on upper extremity functions and trunk control of individuals with cerebral palsy.All individuals diagnosed with Cerebral Palsy who agree to participate in the study and meet the inclusion criteria will be randomly divided into two groups as Study and Control Group. In addition to conventional physiotherapy, the study group will be trained in the Hippotherapy Simulature for 15 minutes a day, 5 days a week for 4 weeks.n addition to conventional physiotherapy, the control group will be allowed to sit in the Hippotherapy Simulature for 15 minutes a day, 5 days a week for 4 weeks. However, the simulator will be kept in closed position to prevent oscillations.

DETAILED DESCRIPTION:
Cerebral Palsy can be defined as a non-progressive lesion that occurs in the brain that has not yet completed its development and causes activity limitation with movement and posture problems. Although the disorders seen in Cerebral Palsy are not progressive, these individuals may experience losses in their current motor functions in later ages and this may cause losses in their independence and activities of daily living. The hippotherapy simulator imitates the three-dimensional mechanical movement and walking of the horse and transfers the mechanical effect to the rider during hippotherapy. The aim of this study was to investigate the effect of exercise program with hippotherapy simulator on upper extremity functions and trunk control of individuals with cerebral palsy.All individuals diagnosed with Cerebral Palsy who agree to participate in the study and meet the inclusion criteria will be randomly divided into two groups as Study and Control Group. In addition to conventional physiotherapy, the study group will be trained in the Hippotherapy Simulature for 15 minutes a day, 5 days a week for 4 weeks.n addition to conventional physiotherapy, the control group will be allowed to sit in the Hippotherapy Simulature for 15 minutes a day, 5 days a week for 4 weeks. However, the simulator will be kept in closed position to prevent oscillations.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6-18 years old
* Being diagnosed with unilateral spastic type cerebral palsy
* Voluntariness of the family and individuals to participate in the study
* Being at I, II, III level according to the Hand Skills Classification System
* To have the cognitive development to cooperate

Exclusion Criteria:

* Having undergone any orthopedic and/or neurological surgery and/or BoNT A operation within the last 6 months
* Having a history of epilepsy
* Hearing and/or vision loss at a level that prevents participation in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Hand Function assessment | 2 minutes
  Jabson Taylor hand function test will be used. The test measures the accuracy of speed and performance on a variety of grip and release tasks using everyday items.

SECONDARY OUTCOMES:
Trunk control assessment | 2 minutes
  The Trunk Control Measurement Scale (TCMS) will be used to assess trunk control in the participants. The fifteen-item SCS assesses static and dynamic components of the trunk during sitting.
Balance assessment | 2 minutes
  Timed up and go test will be used to evaluate balance. The patient is asked to stand up from the chair without support from the chair, walk 3 m, walk back towards the chair without touching anything and take the sitting position again. The time starts when the patient stands up from the chair and ends when the patient returns to the chair and sits down again.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No